CLINICAL TRIAL: NCT00881634
Title: A Single-Dose Comparative Bioavailability Study of Two Formulations of Cetirizine Hydrochloride/Pseudoephedrine Hydrochloride 5 mg/120 mg Extended Release Tablets Under Fed Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Cetirizine Hydrochloride/Pseudoephedrine Hydrochloride 5 mg/120 mg Extended Release (ER) Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2005-984
Record Dates: First submitted 2009-04-13; First posted 2009-04-15 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2009-04

CONDITIONS: Allergies
MeSH Terms: conditions — Hypersensitivity

ARMS (2):
- 1 (Experimental): Cetirizine HCl/Pseudoephedrine HCl 5 mg/120 mg Tablets (Sandoz, USA)
  Interventions: Drug: Cetirizine HCl/Pseudoephedrine HCl 5 mg/120 mg Tablets (Sandoz, USA)
- 2 (Active Comparator): Zyrtec-D 12 Hour 5 mg/120 mg Extended Release Tablets (Pfizer, USA)
  Interventions: Drug: Zyrtec-D 12 Hour 5 mg/120 mg Extended Release Tablets (Pfizer, USA)

INTERVENTIONS:
Drug: Cetirizine HCl/Pseudoephedrine HCl 5 mg/120 mg Tablets (Sandoz, USA)
  Arms: 1
Drug: Zyrtec-D 12 Hour 5 mg/120 mg Extended Release Tablets (Pfizer, USA)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Cetirizine Hydrochloride/Pseudoephedrine Hydrochloride 5 mg/120 mg ER tablets under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 20 Years to 53 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Xueyu (Eric) Chen, M.D., Principal Investigator — Pharma Medica Research, Inc.